CLINICAL TRIAL: NCT05153850
Title: Assessment of the Response to the Complete Vaccination Guidelines Against Sars-cov2 in Patients With Inflammatory Bowel Disease Under Inmunosuppressor Treatment
Brief Title: Assessment of the Response to the Complete Vaccination Guidelines Against Sars-cov2
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-COV-2021-01
Record Dates: First submitted 2021-12-09; First posted 2021-12-10 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients diagnosed with inflammatory bowel disease with the complete vaccination regimen.

SUMMARY:
Prospective observational single-center study in which the impact of anti-TNF biological treatment on the humoral response after complete vaccination against SARS-COV2 in patients with inflammatory bowel disease is analyzed.

DETAILED DESCRIPTION:
Prospective observational single-center study in which the impact of anti-TNF biological treatment on the humoral response after complete vaccination against SARS-COV2 in patients with inflammatory bowel disease is analyzed.

The first objective is to compare the seroconversion rate after full vaccination against SARS-COV2 in patients with IBD treated with anti-TNF drugs versus patients treated with Ustekinumab / Vedolizumab and patients without immunosuppressive treatment.

The Patients included in the study belong to the health area of the Virgen Macarena University Hospital who meet the following inclusion criteria and none for exclusion.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age (> 18 years).
* Diagnosis of inflammatory bowel disease (Crohn's Disease or Ulcerative Colitis).
* Complete vaccination schedule (one or two doses depending on previous SARS-Cov2 infection) between one and four months prior to the determination of anti-SARS-Cov2 antibodies.
* Treatment with biological therapy for at least 6 weeks prior to the time of vaccination for the group of patients treated with biological drugs.

Exclusion Criteria:

* Last vaccination dose more than four months ago from the determination of antibodies against SARS-Cov2.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients included in the study are elderly patients suffering from inflammatory bowel disease and have completed their vaccination schedule against the SARS-COV-2 virus.
Sampling Method: Probability Sample
Enrollment: 243 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with peripheral blood antibodies against SARS-COV2. | Up to 16 weeks.
  Seroconversion rate against SARS-COV2 defined as the presence of antibodies in peripheral blood four months after the complete vaccination schedule against SARS-COV2.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Argüelles Arias, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Andalusia, Spain